CLINICAL TRIAL: NCT00341120
Title: Methylenetetrahydrofolate Reductase C677T Mutation, Other Variant Genotypes, and Male Infertility
Brief Title: Genetic Causes of Male Infertility
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999903076; 03-CH-N076
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2012-08-29

CONDITIONS: Male Infertility
Keywords: Genotypes; Mutation; Folate; Male Infertility; Nutrition
MeSH Terms: conditions — Infertility, Male

SUMMARY:
This study is being conducted at the University Hospital of Lund University in Malmo, Sweden, in collaboration with the U.S. National Institute of Child Health and Human Development. The study will try to identify genetic causes of impaired sperm production and male infertility. It will focus on the possible role of the MTHFR and CBS genes, which regulate absorption and metabolism of the vitamin, folate in infertility. If the nutritional intake or metabolism of this vitamin is related to male infertility, then this cause of infertility would be potentially curable.

Fertile and infertile men between 20 and 45 years of age may be eligible for this study. Criteria include the following:

* Fertile men: men whose partners are younger than age 40 and are attending Lund University prenatal clinic; who have fathered one or more pregnancies and who stopped birth control to achieve the present pregnancy; who achieved the present pregnancy in less than 12 months of unprotected intercourse.
* Infertile men: men referred to the Scandian Andrology Centre whose infertility is unexplained, whose partners are younger than age 40 and who have had regular sexual intercourse without contraception for at least 12 months without achieving a pregnancy.

All participants will have the following tests and procedures:

* Complete a questionnaire providing information about their reproductive and medical history and recent dietary history;
* Provide blood samples for analysis of red cell folate, plasma folate, plasma homocysteine, plasma B12, and for genetic evaluation;
* Provide a semen sample for routine analysis, including volume, sperm concentration, sperm motility, and sperm morphology.

In addition, infertile men will undergo a physical examination and review of their medical records.

DETAILED DESCRIPTION:
It is evident that genetic variation plays a substantial role in the etiology of male infertility. Studies of children fathered through intracytoplasmic sperm injection or ICSI have revealed mutations on the AZF region of the Y chromosome linked to male infertility. Mutations of other genes may also be involved. Candidates would include genes for the androgen receptor, follicle-stimulating hormone, and luteinizing hormone, and genes involved in the regulation of spermatogenesis and sperm motility. Mutations in mitochondrial DNA have been linked to poor sperm motility and raise the possibility that some types of male subfertility may be inherited only through the female line.

We propose to assess the role of folate/homocysteine status and MTHFR and CBS gene variants in infertile men in Sweden with no known cause for their infertility and whose wives/partners appear to be fertile. We propose to perform the study in Sweden since Sweden, unlike the U.S., at present does not mandate the enrichment of flour or other foodstuffs with folate.

ELIGIBILITY:
* INCLUSION CRITERIA INFERTILE MEN:

Referred to the Scanian Andrology Centre.

Age 20-45.

Partner age less than 40.

Having had regular sexual intercourse without contraception for a year or more without achieving a pregnancy.

EXCLUSION CRITERIA INFERTILE MEN:

Klinefelters syndrome.

Hypogondotropic hypogonadism.

Y-chromosome microdeletion or abnormality.

Other genetic cause for infertility.

Obstructive azoospermia.

Partner with salpingitis.

Partner with polycystic ovarian syndrome.

Partner with disturbance of ovulation.

Partner with endometriosis.

History of cancer.

History of treatment with cytotoxic drugs, irradiation, or sulfasalazopyrine.

History of cryptorchidism.

History of mumps orchitis.

History of vasectomy.

INCLUSION CRITERIA FERTILE MEN:

Partner attending Lund University prenatal clinic.

Age 20-45.

Partner age less than 40.

Having fathered one or more pregnancies.

Having stopped birth control to achieve present pregnancy.

Having achieved present pregnancy in less than 12 months of unprotected intercourse.

EXCLUSION CRITERIA FERTILE MEN:

History of cancer.

History of treatment with cytotoxic drugs, irradiation, or sulfasalazopyrine.

History of cryptorchidism.

History of mumps orchitis.

Having sought or partner having sought treatment or investigation for fertility.

Ages: 20 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 400 (Actual)
Dates: Start 2003-01-02; Study Completion 2012-08-29

CONTACTS AND LOCATIONS:
Overall Officials: Richard J Levine, M.D., Principal Investigator — Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD)
Locations (1):
- Malmo University Hospital, Malmo, Sweden

REFERENCES:
- [Background] Ma K, Mallidis C, Bhasin S. The role of Y chromosome deletions in male infertility. Eur J Endocrinol. 2000 May;142(5):418-30. doi: 10.1530/eje.0.1420418. PMID 10802517
- [Background] Ford WC. Biological mechanisms of male infertility. Lancet. 2001 Apr 21;357(9264):1223-4. doi: 10.1016/s0140-6736(00)04452-4. No abstract available. PMID 11418145
- [Background] Ruiz-Pesini E, Lapena AC, Diez-Sanchez C, Perez-Martos A, Montoya J, Alvarez E, Diaz M, Urries A, Montoro L, Lopez-Perez MJ, Enriquez JA. Human mtDNA haplogroups associated with high or reduced spermatozoa motility. Am J Hum Genet. 2000 Sep;67(3):682-96. doi: 10.1086/303040. Epub 2000 Aug 9. PMID 10936107